CLINICAL TRIAL: NCT04025645
Title: Common Bile Duct Pressures in Patients With and Without Cholelithiasis: A Cases and Controls Study
Brief Title: Common Bile Duct Pressures in Patients With and Without Cholelithiasis
Status: Completed | Type: Observational
Sponsor: Hospital de La Serena (Other)
Responsible Party: Principal Investigator, MARCELO BELTRAN, Digestive surgeon, Hospital de La Serena
Other Study IDs: HLS-MBS-001
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Biliary Disease
Keywords: Cholelithiasis; Common Bile Duct; Sphincter of Oddi; Amylase; Lipase
MeSH Terms: conditions — Gallbladder Diseases; Cholelithiasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PATIENTS WITH CHOLELITHIASIS: COMMON BILE DUCT PRESSURES WERE MEASURED IN PATIENTS WITH CHOLELITHIASIS
  Interventions: Diagnostic Test: MEASUREMENT OF COMMON BILE DUCT PRESSURES
- PATIENTS WITHOUT CHOLELITHIASIS: COMMON BILE DUCT PRESSURES WERE MEASURED IN PATIENTS WITHOUT CHOLELITHIASIS
  Interventions: Diagnostic Test: MEASUREMENT OF COMMON BILE DUCT PRESSURES

INTERVENTIONS:
Diagnostic Test: MEASUREMENT OF COMMON BILE DUCT PRESSURES — THE PRESSURES OF THE COMMON BILE DUCT WERE MEASURED

SUMMARY:
Objective. To measure the pressures of the common bile duct in patients with and without cholelithiasis and relating them to the presence of pancreatobiliary reflux.

Summary Background Data. The reflux of pancreatic enzymes into the epithelium of the bile duct and mainly of the gallbladder is an abnormal phenomenon that plays a role in the lithogenesis and carcinogenesis of this epithelium. It has been suggested that the cause of this reflux is the dysfunction of the sphincter of Oddi. Because the pressure of the common bile duct depends on the pressures of the sphincter of Oddi, this dysfunction would be reflected in an increase in the pressure of the common bile duct in patients with cholelithiasis.

Methods. A prospective case-control study was designed. The universe was constituted by a convenience sample in which all patients undergoing gastrectomy for gastric cancer during 30 months in our institution were included. The primary outcome measure was to establish differences between common bile duct pressures in patients with and without cholelithiasis.

Results. Common bile duct pressures in patients with gallstones showed a significant elevation (Mean 16.9 mmHg) compared to those of patients without gallstones (Mean 3.3 mm Hg) (p<0.0001). These pressures correlated with the values of amylase and lipase in gallbladder bile; higher levels of these enzymes were found in patients with gallstones compared to patients without gallstones (p<0.0001).

Conclusions. Common bile duct pressures in patients with cholelithiasis were significantly elevated above the parameters previously considered normal.

DETAILED DESCRIPTION:
A prospective study of cases and controls was designed using a previously validated model for the study of occult pancreatobiliary reflux in patients undergoing gastrectomy for gastric cancer, in which cholecystectomy is routine according to the oncological surgery protocol for gastric cancer of our institution. The study universe was constituted by a convenience sample in which all patients undergoing gastrectomy for gastric cancer during the period between January 2015 and June 2017 the investigators included. All patients included in this study signed a detailed informed consent regarding the interventions to be performed and the objectives of the study.

Cholecystectomy was performed in all patients after the section of the duodenum. Before the manipulation and dissection of the Calot triangle, a sample of 5 to 10 cc of bile was taken directly from the gallbladder. The sample was stored in a sterile tube at room temperature and immediately sent for processing. The technicians of our institutional laboratory that processed the sample did not know the details of the study. The cholecystectomy was then carried out until the cystic was reached and was cut as proximally as possible to the gallbladder. Through the cystic duct, a 4 French feeding tube equivalent to 1.35 mm in diameter (Well Lead®, Hamburg, Germany) was introduced until reaching a distance of 3 cm distal to the junction of the cystic duct and the common bile duct. Once tested for patency, this probe was connected to a standard pressure transducer used to measure intra-arterial pressure (Edwards Lifesciences™, Irvine, California, USA) and this was connected to a B40 monitor (General Electric® Medical Systems, Milwaukee, WI, USA) with the ability, among other functions, to perform pressure measurements in millimeters of mercury. The level of the junction of the cystic duct and the common bile duct was taken as a zero point, as previously described. Once the whole system was irrigated with 0.9% physiological solution and the zero point was established on the monitor with the system closed, the system was opened and pressures were measured. The minimum, maximum and mean pressures were recorded for one minute. After the procedure was completed, the gastrectomy was performed.

ELIGIBILITY:
Inclusion Criteria:

* All patients with normal values of amylase, lipase, and liver function tests measured 24 hours before the intervention

Exclusion Criteria:

* Patients previously cholecystectomized
* Patients with clinical, radiological and laboratory evidence of common bile duct stones

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with gastric cancer undergoing elective surgery
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
Common bile duct pressures | Two and a half years
  Establish differences between common bile duct pressures in patients with and without gallstones

SECONDARY OUTCOMES:
Levels of amylase and lipase in bile | Two and a half years
  Establish the relationship between these pressure differences and the presence of pancreatobiliary reflux in patients with and without cholelithiasis

IPD SHARING:
Plan to Share IPD: No